CLINICAL TRIAL: NCT04955691
Title: Metabolic and Neurological Changes Induced by a Very Low Carbohydrate Diet in Youth With Type 1 Diabetes
Brief Title: Metabolic Changes Induced by a Very Low Carbohydrate Diet in Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2000029479; 1K23DK128560-01 (NIH); 2P30DK045735-26 (NIH)
Record Dates: First submitted 2021-07-01; First posted 2021-07-09 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Type1diabetes, Low Carbohydrate Diet
MeSH Terms: interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low carbohydrate diet (Experimental): In this crossover study, participants will be randomized to either a low or standard carbohydrate for 2 weeks. Participants in the low carbohydrate group will limit carbohydrate intake to 15% of total daily calories.
  Interventions: Other: low carbohydrate diet
- standard carbohydrate diet (Active Comparator): In this crossover study, participants will be randomized to either a low or standard carbohydrate for 2 weeks. Participants in the standard carbohydrate group will follow an ad libitum diet with standard carbohydrate intake.
  Interventions: Other: standard carbohydrate diet

INTERVENTIONS:
Other: low carbohydrate diet — Participants will engage in a diet that limits carbohydrate intake to 15% of total daily calories for 2 weeks.
  Arms: low carbohydrate diet
Other: standard carbohydrate diet — Participants will engage in a diet that recommends standard carbohydrate intake with respect to total daily calories for 2 weeks.
  Arms: standard carbohydrate diet

SUMMARY:
As more adolescents with type 1 diabetes (T1D) opt to follow very low carbohydrate diets to improve glucose control, it is becoming increasingly important to study the metabolic and neurological changes that occur on these diets and how these effect patient safety. Understanding the impact of dietary changes on metabolic and neurological factors will help guide clinical advice about the overall safety and efficacy of these diets in the pediatric T1D population. This work will be the basis of future studies testing dietary interventions to improve glycemic control and ensure that these dietary interventions are safe for growing youth with T1D.

DETAILED DESCRIPTION:
The primary objective of this randomized crossover study is to determine whether a very low carbohydrate diet improves glycemic changes (measured by continuous glucose monitors) when compared to a standard carbohydrate diet in youth with type 1 diabetes.

The secondary objectives of the study are to compare metabolic changes after 2 weeks on each diet using the 2-step hyperinsulinemic euglycemic-hypoglycemic clamp and stable isotope infusions. The euglycemic portion of the clamp will allow us to determine the hepatic glucose production and adipose tissue lipolysis. Secondary objectives also include measuring the neurohormonal response to hypoglycemia after 2 weeks on each diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes for at least 1 year
* Hemoglobin A1c level < 10% within the past 2 months
* Provision of signed and dated informed consent form by the adult (if person is at least 18 years old) or parent and assent form if the participant is <18 years old.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* All sexes are eligible
* Diagnosis of type 1 diabetes for at least 1 year
* Insulin pump use for at least 2 months.
* Ability to perform daily blood ketone checks, wear a continuous glucose monitor, willing to wear an activity monitor, willing to adhere to the study diets and keep a diet journal.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of the dietary intervention.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

* Current use of glucose-lowering agents other than insulin
* Unstable psychiatric disorders, including eating disorders
* Weight loss medications within the last 6 months
* Pregnancy or lactation, or planning pregnancy within the next 6 months
* BMI < 19 kg/m2 for individuals 18 years of age or older
* BMI < 5%ile for individuals under 18 years
* Weight less than 49 kg or 108 pounds
* Other medical conditions that may interfere with glucose metabolism and insulin sensitivity

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Nally, M.D., Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Carbohydrate Diet, Then Standard Carbohydrate Diet: In this crossover study, participants will be randomized to either a low or standard carbohydrate for 2 weeks. Participants in the low carbohydrate group will limit carbohydrate intake to 15% of total daily calories.
  low carbohydrate diet: Participants will engage in a diet that limits carbohydrate intake to 15% of total daily calories for 2 weeks.
- Standard Carbohydrate Diet, Then Low Carbohydrate Diet: In this crossover study, participants will be randomized to either a low or standard carbohydrate for 2 weeks. Participants in the standard carbohydrate group will follow an ad libitum diet with standard carbohydrate intake.
  standard carbohydrate diet: Participants will engage in a diet that recommends standard carbohydrate intake with respect to total daily calories for 2 weeks.
Period: Period 1
Arm/Group | Low Carbohydrate Diet, Then Standard Carbohydrate Diet | Standard Carbohydrate Diet, Then Low Carbohydrate Diet
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Washout
Arm/Group | Low Carbohydrate Diet, Then Standard Carbohydrate Diet | Standard Carbohydrate Diet, Then Low Carbohydrate Diet
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Low Carbohydrate Diet, Then Standard Carbohydrate Diet | Standard Carbohydrate Diet, Then Low Carbohydrate Diet
Started | 9 | 10
Analyzed | 9 | 10
Completed | 8 | 8
Not Completed | 1 | 2
Not completed — Discontinued intervention | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Carbohydrate Diet, Then Standard Carbohydrate Diet | Standard Carbohydrate Diet, Then Low Carbohydrate Diet | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (3) | 17 (2.67) | 17 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 8 | 7 | 15
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percent Time in the Optimal Glucose Range
Description: Time in the optimal glucose range will be operationally defined as the percent time spent in the target range of 70-180 mg/dL during the 2 weeks.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet
Number analyzed (Participants) | 19 | 19
percentage of time | 71.20 [68.53 to 73.87] | 62.51 [59.82 to 65.20]
Statistical Analysis 1: Comparison: Low Carbohydrate Diet; Test type: Superiority; p < 0.001, t-test, 1 sided

2. Secondary Outcome: Percent Time Spent With Hypoglycemia.
Description: Time spent with hypoglycemia will be operationally defined as the percent time spent in the hypoglycemic ranges during 2 weeks of diet. Level 2 hypoglycemia defined as <54 mg/dL. Level 1 hypoglycemia defined as 54-69 mg/dL.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet
Number analyzed (Participants) | 19 | 19
percentage of time
  <54 mg/dL | 0.42 [0.15 to 0.69] | 0.33 [0.20 to 0.45]
  54-69 mg/dL | 1.27 [0.91 to 1.62] | 1.46 [1.15 to 1.77]
Statistical Analysis 1: Comparison: Low Carbohydrate Diet vs Standard Carbohydrate Diet; <54 mg/dL; Test type: Superiority; p = 0.57, t-test, 1 sided
Statistical Analysis 2: Comparison: Low Carbohydrate Diet vs Standard Carbohydrate Diet; 54-69 mg/dL; Test type: Superiority; p = 0.43, t-test, 1 sided

3. Secondary Outcome: Percent Time Spent With Hyperglycemia
Description: Time spent with hyperglycemia will be operationally defined as the percent time spent in the hyperglycemic ranges during 2 weeks of diet. Level 1 hyperglycemia defined as 181-250 mg/dL. Level 2 hyperglycemia defined as >250 mg/dL.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet
Number analyzed (Participants) | 19 | 19
percentage of time
  181-250 mg/dL | 19.93 [18.23 to 21.63] | 23.20 [21.59 to 24.82]
  >250 mg/dL | 7.19 [5.7 to 8.67] | 12.5 [10.57 to 14.43]
Statistical Analysis 1: Comparison: Low Carbohydrate Diet vs Standard Carbohydrate Diet; 181-250 mg/dL; Test type: Superiority; p = 0.006, t-test, 1 sided
Statistical Analysis 2: Comparison: Low Carbohydrate Diet vs Standard Carbohydrate Diet; >250 mg/dL; Test type: Superiority; p < 0.001, t-test, 1 sided

4. Other Pre Specified Outcome: Human Factors
Description: To describe how participants feel about and react to following a very low carbohydrate diet, interviews will be conducted. Data will be coded and emerging patterns will be combined into descriptive themes.
Time Frame: 8 weeeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Washout Period: Washout period between the 2 diets
Arm/Group | Low Carbohydrate Diet | Standard Carbohydrate Diet | Washout Period
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 8/19 | 8/19 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Carbohydrate Diet (N=19) | Standard Carbohydrate Diet (N=19) | Washout Period (N=19)
Nausea/Vomiting with elevated ketone levels (General disorders) | 2 | 0 | 0
Elevated ketone levels without symptoms (General disorders) | 2 | 1 | 0
Infusion site failure with elevated ketones (Injury, poisoning and procedural complications) | 1 | 1 | 0
Infusion site failure with hyperglycemia (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Pain at intravenous site (Injury, poisoning and procedural complications) | 1 | 2 | 0
Viral illness with vomiting (General disorders) | 1 | 0 | 0
Hypoglycemia during clamp (Endocrine disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Allergic reaction to cough syrup (General disorders) | 0 | 1 | 0
ER visit for foot pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Allergic reaction to fitness tracker wrist band (General disorders) | 0 | 1 | 0
ER visit for foot injury (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT04955691/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04955691/ICF_001.pdf